CLINICAL TRIAL: NCT06508424
Title: Investigating the Glycaemic and Satiating Capacity of PulseOn® Enriched Foods: a Randomised Control Trial
Brief Title: Investigating the Glycaemic and Satiating Capacity of PulseOn® Enriched Foods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Quadram Institute Bioscience (Other); Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Principal Investigator, Anna Sorsby, Senior Lecturer in Nutrition, Sheffield Hallam University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ER64439232
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Glycaemic Response; Appetitive Behavior; Energy Intake
MeSH Terms: conditions — Appetitive Behavior | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the treatment (PulseOn) or control group at the outset of their participation. Following a minimum of a one-week washout period, participants will then participate in the alternative arm.
Who Masked: Participant
Masking Description: Participants will not be told which arm of the trial they are taking part in. PulseOn crackers and the wheat flour control crackers have been matched as closely as possible for energy content and sensory characteristics. Participants will be asked to rate the acceptability of the crackers to determine whether there are any discernible differences, however they are required to consume a set amount.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PulseOn enriched crackers (Experimental): PulseOn enriched crackers
  Interventions: Other: PulseOn
- Wheat Flour Control (Placebo Comparator): Wheat Flour Control
  Interventions: Other: Wheat flour control

INTERVENTIONS:
Other: PulseOn — PulseOn - 1 week washout period between interventions 75g crackers
  Arms: PulseOn enriched crackers
Other: Wheat flour control — Control -1 week washout period between interventions 75g crackers
  Other Names: Wheat flour
  Arms: Wheat Flour Control

SUMMARY:
The purpose of this randomised control trial is to determine whether consuming PulseOn enriched crackers for breakfast influences post-prandial glycaemic response and markers of appetite (hunger, fullness, desire to eat) over 4 hours, and energy intake at an ad libitum lunch meal on the same day. Healthy individuals with no underlying metabolic disease will be recruited to take part in this study.

DETAILED DESCRIPTION:
PulseON® is a unique flour that is made 100% from pulses, but unlike other flours it has been obtained through an alternative milling process (WO2019155190) which preserves whole plant cells (Edwards et al., 2020). These cells were shown to remain intact during down-stream processing into food products including bread and biscuits, and influence glycaemic response to these foods (Delamare et al., 2020; Bajka et al., 2021). Interestingly, the PulseON®-enriched breads also significantly enhanced and prolonged release of the gut hormones glucagon-like peptide-1 (GLP1) and peptide YY (PYY), which are known to have anorexigenic effects (Bajka et al., 2023). Studies using chick pea purees and hummus products have also shown positive findings in relation to appetite sensations and food intake (Pälchen et al., 2022; Alshaalan et al., 2024).

This work aims to recruit 50 participants through the use of posters and emails at Sheffield Hallam University, as well as in the local Sheffield area and through social media.

-30 minutes - baseline measures (body mass index (kg/m2), waist circumference (cm), blood glucose (mmol/l), hunger, fullness, desire to eat) are taken

0 minutes - pre-load consumed within 15 minutes (75g wheat flour / PulseOn crackers) The wheat flour cracker is made from 100% wheat flour. The PulseOn cracker is made from 40% PulseOn flour and 60% wheat flour.

30, 45, 60, 75, 90, 105, 120, 150, 180, 210 minutes - repeat baseline measures

240 minutes - ad libitum lunch provided (pasta and tomato sauce) and participants instructed to eat to fullness.

Paired sample t-tests will be used to compare measures between the two visits.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18y

Exclusion Criteria:

* smoker / recreational drug user
* restrained eater (as determined by the three factor eating questionnaire (TFEQ-R18))
* vegan
* pregnant / lactating
* blood clotting disorder
* taking medication for heart / metabolic disease
* pacemaker fitted
* energy restricted diet or lost >5% body weight in the last 3 months
* elite athletes
* dysphagia
* food allergy / intolerance
* disease / inflammation of the GI tract

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Energy Intake at a test meal | Participants consume the preload at 0 minutes, and the test meal at 240mins.
  Following the consumption of either the control / PulseOn enriched preload (crackers), participants will be asked to consume a standardised lunch meal of pasta and tomato sauce until they are full. The amount consumed will be measured using the Sussex Ingestion Pattern Monitor, and reported in grams and kcals.
Glycaemic response | Baseline blood measures to be taken at -30 minutes. Participants consume the preload at 0 minutes, and capillary blood samples are measured at 30, 45, 60, 75, 90, 105, 120, 150, 180 and 210 minutes.
  Following the consumption of either the control / PulseOn enriched preload (crackers), capillary blood samples will be measured at 15 / 30 minute intervals up to lunch time.
Markers of appetite | Baseline hunger, fullness and desire to eat to be taken at -30 minutes. Participants consume the preload at 0 minutes, and further hunger, fullness and desire to eat measures are taken at 30, 45, 60, 75, 90, 105, 120, 150, 180 and 210 minutes.
  Following the consumption of either the control / PulseOn enriched preload (crackers), hunger, fullness and desire to eat will be measured at 15 / 30 minute intervals up to lunch time using visual analogue scale.

SECONDARY OUTCOMES:
Mood | Baseline mood ratings will be measured at -30 minutes. Participants consume the preload at 0 minutes, and further mood ratings are measured at 30, 45, 60, 75, 90, 105, 120, 150, 180 and 210 minutes.
  Following the consumption of either the control / PulseOn enriched preload (crackers), the following attributes will be measured at 15 / 30 minute intervals up to lunch time using visual analogue scale - happy, relaxed, energetic, thirsty, nauseous.
Post intervention food / energy / nutrient intake | 24hrs post intervention
  Following the completion of the lab-based study, participants will leave the research facility and complete a 24hr estimated measures diet diary which will be analysed on Nutritics.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline E Millman, PhD, Principal Investigator — Sheffield Hallam University
Locations (1):
- Food and Nutrition Group, Sheffield Hallam University, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edwards, C. H., Ryden, P., Pinto, A. M., van Der Schoot, A., Stocchi, C., Perez-Moral, N., ... & Ellis, P. R. (2020). Chemical, physical and glycaemic characterisation of PulseON®: A novel legume cell-powder ingredient for use in the design of functional foods. Journal of Functional Foods, 68, 103918.
- [Background] Delamare GYF, Butterworth PJ, Ellis PR, Hill S, Warren FJ, Edwards CH. Incorporation of a novel leguminous ingredient into savoury biscuits reduces their starch digestibility: Implications for lowering the Glycaemic Index of cereal products. Food Chem X. 2020 Feb 7;5:100078. doi: 10.1016/j.fochx.2020.100078. eCollection 2020 Mar 30. PMID 32140680
- [Background] Bajka BH, Pinto AM, Ahn-Jarvis J, Ryden P, Perez-Moral N, van der Schoot A, Stocchi C, Bland C, Berry SE, Ellis PR, Edwards CH. The impact of replacing wheat flour with cellular legume powder on starch bioaccessibility, glycaemic response and bread roll quality: A double-blind randomised controlled trial in healthy participants. Food Hydrocoll. 2021 May;114:106565. doi: 10.1016/j.foodhyd.2020.106565. PMID 33941996
- [Background] Bajka BH, Pinto AM, Perez-Moral N, Saha S, Ryden P, Ahn-Jarvis J, van der Schoot A, Bland C, Berry SE, Ellis PR, Edwards CH. Enhanced secretion of satiety-promoting gut hormones in healthy humans after consumption of white bread enriched with cellular chickpea flour: A randomized crossover study. Am J Clin Nutr. 2023 Mar;117(3):477-489. doi: 10.1016/j.ajcnut.2022.12.008. Epub 2022 Dec 28. PMID 36811474
- [Background] Palchen K, Bredie WLP, Duijsens D, Isaac Alfie Castillo A, Hendrickx M, Van Loey A, Raben A, Grauwet T. Effect of processing and microstructural properties of chickpea-flours on in vitro digestion and appetite sensations. Food Res Int. 2022 Jul;157:111245. doi: 10.1016/j.foodres.2022.111245. Epub 2022 Apr 12. PMID 35761557
- [Background] Alshaalan RA, Charalambides MN, Edwards CH, Ellis PR, Alrabeah SH, Frost GS. Impact of chickpea hummus on postprandial blood glucose, insulin and gut hormones in healthy humans combined with mechanistic studies of food structure, rheology and digestion kinetics. Food Res Int. 2024 Jul;188:114517. doi: 10.1016/j.foodres.2024.114517. Epub 2024 May 10. PMID 38823849